CLINICAL TRIAL: NCT06548347
Title: A International Multicenter, Randomized, Double-Blind, Controlled Phase II/III Study to Evaluate the Efficacy and Safety of Linperlisib Plus CHOP Versus CHOP in Patients With Newly Diagnosed Peripheral T Cell Lymphoma
Brief Title: A Phase II/III Study of Linperlisib Plus CHOP Versus CHOP in Patients With Newly Diagnosed Peripheral T Cell Lymphoma
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai YingLi Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YY-20394-015
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Linperlisib80mg+CHOP (Experimental)
  Interventions: Drug: Linperlisib
- Linperlisib60mg+CHOP (Experimental)
  Interventions: Drug: Linperlisib
- CHOP (Active Comparator)
  Interventions: Drug: Linperlisib

INTERVENTIONS:
Drug: Linperlisib — Linperlisib at 80 mg orally once daily (QD) or 60mg orally once daily (QD) plus CHOP, placebo at 80mg or 60 mg orally once daily (QD) plus CHOP for 6 cycles
  Other Names: CHOP

SUMMARY:
This is a Phase II/III, international multiple center study to evaluate the efficacy, safety, and PK of Linperlisib plus CHOP and CHOP in adult patients with Newly Diagnosed Peripheral T Cell Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult patient 18-70 years of age at the time of signing the informed consent.

  2. Diagnosis of one of the following histologic subtypes of PTCL, pathologically confirmed, as defined by the WHO 2017 classification system:
  1. Peripheral T-cell lymphoma-not otherwise specified (PTCL-NOS)
  2. Angioimmunoblastic T-cell lymphomas (AITL)
  3. Anaplastic large cell lymphoma (ALCL). ALK positive or ALK negative
  4. Monomorphic epitheliotropic intestinal T-cell lymphoma (MEITL).
  5. Follicular T-cell Lymphoma (FTCL). 3. Newly diagnosed and has no received systemic therapy for PTCL. 4. Has a life expectancy ≥6 months. 5. For patients with CD30+ PTCL, progressed on or are ineligible or intolerant to brentuximab vedotin, or progressed on or are ineligible or intolerant to regional standard of care if brentuximab vedotin not approved or not available.

     6. Agree to provide archival tumor tissue samples or undergo pretreatment fresh tissue biopsy.

     7. Has radiographically measurable disease of PTCL as per Lugano Criteria with at least one measurable disease lesion > 1.5 cm in at least one dimension (which has not been previous radiated) by 18FDG-PET-CT, MRI, or diagnostic CT within 28 days prior to start of study treatment.

     8. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.

     9. Has adequate organ function as defined below: System Laboratory Value Haematological Absolute neutrophil count ≥1.5×109/L Note: No growth factor supports within 14 days of first dose Platelet count ≥75×109/L Note: No blood product transfusion is allowed within 14 days of first dose Haemoglobin ≥80 g/L Note: criteria must be met without erythropoietin dependency and no blood product transfusion is allowed within 14 days of first dose Hepatic Total bilirubin ≤1.5×ULN Note: Patients with Gilbert's Syndrome or other benign congenital hyperbilirubinemia may be eligible at the Investigator's discretion in consultation with the Medical Monitor, if ≤ 3 × ULN Alanine aminotransferase ≤2.5×ULN Note: ≤ 5 × ULN if there is liver involvement by lymphoma Aspartate aminotransferase ≤2.5×ULN Note: ≤ 5 × ULN if there is liver involvement by lymphoma Renal CrCl calculated by Cockcroft-Gault formula CrCl ≥50 mL/min or SCr≤1.5×ULN Cardiac Left ventricular ejection fraction LVEF ≥ 50% by an echocardiogram (ECHO) or multigated acquisition scan (MUGA).

     QTcF <450 ms Abbreviations: CrCl=creatinine clearance; RBC=red blood cell; QTcF=QT interval corrected using Fridericia's formula; ULN=upper limit of normal.

     10. Male patients are eligible to participate if they agree to use a highly effective contraception during the treatment period and for at least 6 months after the last dose of study treatment and refrain from donating sperm during this period 11. Female patients are eligible to participate if they are not pregnant, not breastfeeding, and at least one of the following conditions applies: 12. Patient must be willing and able to adhere to the study and are capable of giving signed informed consent.

     Exclusion Criteria:
* Patients are excluded from the study if any of the following criteria apply:

  1. Has received anti-lymphoma therapy.
  2. Patients with extranodal NK/T-cell lymphoma or CTCL.
  3. Has dropsy of serous cavity not under controlled by surgical drains or other therapy.
  4. Patients with peripheral T-cell lymphoma having known central nervous system (CNS) invasion (either CNS lymphoma or leptomeningeal lymphoma).
  5. Has received systemic steroids (in dosing exceeding 20 mg daily of prednisone equivalent) within 14 days of the first dose of study treatment.
  6. Presence of multiple factors affecting drug administration and absorption such as inability to swallow, diarrhea of CTCAE Grade >1, and ileus. Use of any drug that may result in QT prolongation (e.g., antiarrhythmic agents) cannot be interrupted during the study.
  7. Has a history of or concurrent interstitial lung disease of any severity and/or severely impaired lung function.
  8. Has active viral, bacterial, fungal infection or other serious infection requiring systemic treatment within 14 days before the first dose of study treatment. Routine antimicrobial prophylaxis is permitted.
  9. Has received a live vaccination within 30 days before the first dose of study treatment or is scheduled to be administered during the study period. Examples of live vaccines include but are not limited to the following: measles, mumps, rubella, varicella/zoster, yellow fever, Bacille Calmette-Guérin (BCG) and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
  10. Medical history of other primary malignant tumors in the past 5 years, or any evidence of residual disease from a previously diagnosed malignancy.

      Note: Exceptions are patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (e.g., breast, cervical cancer in situ, superficial bladder tumors [Ta and Tis; carcinoma in situ]) who have undergone curative therapy with no evidence of recurrence, localized prostate cancer previously fully resected undergoing surveillance or other adequately treated Stage 1 cancer currently in complete remission.
  11. Uncontrolled pulmonary fibrosis, acute lung disease, interstitial lung disease, etc;
  12. Has clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (New York Heart Association Classification Class ≥II), or serious cardiac arrhythmia requiring medication, any other cardiac disorder not suitable for participation in this study based on the judgment of the investigator.

      Note: During the treatment period, patients should not take medication that may prolong the QT (such as antiarrhythmic drugs).
  13. Decompensated cirrhosis (Child-Pugh: B or C). Patients with active viral (any etiology) hepatitis (HbsAg and/or HbcAb positive and HBV-DNA positive) are excluded. Patients with a history of hepatitis C virus (HCV) infection (Hepatitis C antibody positive and HCV-RNA positive).
  14. Medical history of immunodeficiency syndrome (AIDS)-defining illness, including Human immunodeficiency virus (HIV) infection, or allogeneic bone marrow/stem cells transplant or organ transplant, or has active autoimmune diseases or has medical history of autoimmune diseases (such as autoimmune enteritis, systemic lupus erythematosus);
  15. Has undergone major surgery (excluding lymph node biopsy) or significant trauma ≤4 weeks before the first dose of study treatment.

      Note: patients must have recovered adequately from surgery prior to starting study treatment.
  16. Has a history or current evidence of any condition, laboratory abnormality or other circumstances that might confound the results of the study or interfere with participation for the full duration of the study, such that it is not in the best interests of the patient to take part in the study.
  17. Medical history of active bleeding within 2 months prior to study entry, or susceptible to bleeding by the judgement of investigator.
  18. Has a history of hypersensitivity to Linperlisib and CHOP and/or any excipients.
  19. Female patient are pregnant, and are breastfeeding.
  20. Has had received prior systemic cytotoxic anticancer therapy, or definitive radiotherapy within 28 days prior to the first dose of study treatment.
  21. Judgment by the investigator that the volunteer should not participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Study treatment will continue until unacceptable toxicity or documented disease progression, or for 2 years, whichever is earlier.
progression-free survival | Study treatment will continue until unacceptable toxicity or documented disease progression, or for 2 years, whichever is earlier.